CLINICAL TRIAL: NCT03661658
Title: Inferior Alveolar Nerve Lateralization With Simultaneous Implant Placement Versus the Use of Short Dental Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ehab Ahmed Shams, dentist-Master student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cairo university 8
Record Dates: First submitted 2018-09-02; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Primary Stability of the Implants; Marginal Bone Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inferior alveolar nerve lateralization with implant placement (Active Comparator)
  Interventions: Procedure: Inferior alveolar nerve lateralization with simultaneous implant placement
- Using short dental implant with atrophic mandible (Experimental)
  Interventions: Procedure: Using short dental implant

INTERVENTIONS:
Procedure: Using short dental implant — Using short dental implant for patients with atrophic posterior mandible.
  Arms: Using short dental implant with atrophic mandible
Procedure: Inferior alveolar nerve lateralization with simultaneous implant placement — Inferior alveolar nerve lateralization with simultaneous implant placement in atrophic posterior mandible.
  Arms: Inferior alveolar nerve lateralization with implant placement

SUMMARY:
Assess the long term stability of short dental implants in comparison to standard implants inserted simultaneously with inferior alveolar nerve lateralization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with edentulous posterior mandible.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.
* Residual alveolar bone width longer than 6 mm height (7-9 mm).

Exclusion Criteria:

* Presence of fenestrations or dehiscence of the residual ridge.
* Heavy smokers more than 20 cigarettes per day .(24)
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Primary stability | 3 months
  measuring the primary stability using the osstel

SECONDARY OUTCOMES:
Marginal bone loss | 3 months
  measuring the marginal bone loss by using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab Ahmed Shams, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes